CLINICAL TRIAL: NCT02792595
Title: Sun Protection Factor Determination (In Vivo Determination of the Sun Protection Factor ISO 24444) (61-SPF-iM)
Brief Title: In Vivo Sun Protection Factor Determination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 204736
Record Dates: First submitted 2015-06-25; First posted 2016-06-07 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Negative Control (Sham Comparator): Untreated area will be irradiated using a sun simulator with UV irradiation increment of 1.25 to detect MED of the unprotected skin.
  Interventions: Other: Negative Control
- Positive Control (Active Comparator): After irradiation of the test area with a sun simulator with an increment of UV radiation of 1.25, positive control will be applied. The dose of positive control will be measured in accordance to the application volume (2 milligram (mg)/centimeter (cm)^2 (± 0.05 mg/cm^2) and it will be applied using a micro litre syringe in approximately 15-30 small droplets all over the test area. Positive control will be then quickly spread by gently rubbing with a non-saturated finger cot, first with rotating followed by crosswise movements for a final uniform coating on the skin. Spreading time will be between 20 and 50 seconds (s). After waiting for 15 to 30 minutes (min), the test area will be again irradiated (increment of 1.12 or 1.25) with the sun simulator. The irradiation time will depend on the SPF of positive control, participants' skin prototype, determined MED after irradiation and actual power of sun simulator.
  Interventions: Other: Positive Control
- Test Product A (Experimental): After irradiation of the test area with a sun simulator with an increment of UV radiation of 1.25, test product will be applied. The dose of test product will be measured in accordance to the application volume (2 mg/cm^2 (± 0.05 mg/cm^2) and it will be applied using a micro litre syringe in approximately 15-30 small droplets all over the test area. Test product will be then quickly spread by gently rubbing with a non-saturated finger cot, first with rotating followed by crosswise movements for a final uniform coating on the skin. Spreading time will be between 20 and 50 s. After waiting for 15 to 30 min, the test area will be again irradiated (increment of 1.12 or 1.25) with the sun simulator. The irradiation time will depend on the expected SPF of the test product, participants' skin prototype, determined MED after irradiation and actual power of sun simulator.
  Interventions: Other: Test Product A
- Test Product B (Experimental): After irradiation of the test area with a sun simulator with an increment of UV radiation of 1.25, test product will be applied. The dose of test product will be measured in accordance to the application volume (2 mg/cm^2 (± 0.05 mg/cm^2) and it will be applied using a micro litre syringe in approximately 15-30 small droplets all over the test area. Test product will be then quickly spread by gently rubbing with a non-saturated finger cot, first with rotating followed by crosswise movements for a final uniform coating on the skin. Spreading time will be between 20 and 50 s. After waiting for 15 to 30 min, the test area will be again irradiated (increment of 1.12 or 1.25) with the sun simulator. The irradiation time will depend on the expected SPF of the test product, participants' skin prototype, determined MED after irradiation and actual power of sun simulator.
  Interventions: Other: Test Product B
- Test Product C (Experimental): After irradiation of the test area with a sun simulator with an increment of UV radiation of 1.25, test product will be applied. The dose of test product will be measured in accordance to the application volume (2 mg/cm^2 (± 0.05 mg/cm^2) and it will be applied using a micro litre syringe in approximately 15-30 small droplets all over the test area. Test product will be then quickly spread by gently rubbing with a non-saturated finger cot, first with rotating followed by crosswise movements for a final uniform coating on the skin. Spreading time will be between 20 and 50 s. After waiting for 15 to 30 min, the test area will be again irradiated (increment of 1.12 or 1.25) with the sun simulator. The irradiation time will depend on the expected SPF of the test product, participants' skin prototype, determined MED after irradiation and actual power of sun simulator.
  Interventions: Other: Test Product C
- Test Product D (Experimental): After irradiation of the test area with a sun simulator with an increment of UV radiation of 1.25, test product will be applied. The dose of test product will be measured in accordance to the application volume (2 mg/cm^2 (± 0.05 mg/cm^2) and it will be applied using a micro litre syringe in approximately 15-30 small droplets all over the test area. Test product will be then quickly spread by gently rubbing with a non-saturated finger cot, first with rotating followed by crosswise movements for a final uniform coating on the skin. Spreading time will be between 20 and 50 s. After waiting for 15 to 30 min, the test area will be again irradiated (increment of 1.12 or 1.25) with the sun simulator. The irradiation time will depend on the expected SPF of the test product, participants' skin prototype, determined MED after irradiation and actual power of sun simulator.
  Interventions: Other: Test Product D
- Test Product E (Experimental): After irradiation of the test area with a sun simulator with an increment of UV radiation of 1.25, test product will be applied. The dose of test product will be measured in accordance to the application volume (2 mg/cm^2 (± 0.05 mg/cm^2) and it will be applied using a micro litre syringe in approximately 15-30 small droplets all over the test area. Test product will be then quickly spread by gently rubbing with a non-saturated finger cot, first with rotating followed by crosswise movements for a final uniform coating on the skin. Spreading time will be between 20 and 50 s. After waiting for 15 to 30 min, the test area will be again irradiated (increment of 1.12 or 1.25) with the sun simulator. The irradiation time will depend on the expected SPF of the test product, participants' skin prototype, determined MED after irradiation and actual power of sun simulator.
  Interventions: Other: Test Product E
- Test Product F (Experimental): After irradiation of the test area with a sun simulator with an increment of UV radiation of 1.25, test product will be applied. The dose of test product will be measured in accordance to the application volume (2 mg/cm^2 (± 0.05 mg/cm^2) and it will be applied using a micro litre syringe in approximately 15-30 small droplets all over the test area. Test product will be then quickly spread by gently rubbing with a non-saturated finger cot, first with rotating followed by crosswise movements for a final uniform coating on the skin. Spreading time will be between 20 and 50 s. After waiting for 15 to 30 min, the test area will be again irradiated (increment of 1.12 or 1.25) with the sun simulator. The irradiation time will depend on the expected SPF of the test product, participants' skin prototype, determined MED after irradiation and actual power of sun simulator.
  Interventions: Other: Test Product F
- Test Product G (Experimental): After irradiation of the test area with a sun simulator with an increment of UV radiation of 1.25, test product will be applied. The dose of test product will be measured in accordance to the application volume (2 mg/cm^2 (± 0.05 mg/cm^2) and it will be applied using a micro litre syringe in approximately 15-30 small droplets all over the test area. Test product will be then quickly spread by gently rubbing with a non-saturated finger cot, first with rotating followed by crosswise movements for a final uniform coating on the skin. Spreading time will be between 20 and 50 s. After waiting for 15 to 30 min, the test area will be again irradiated (increment of 1.12 or 1.25) with the sun simulator. The irradiation time will depend on the expected SPF of the test product, participants' skin prototype, determined MED after irradiation and actual power of sun simulator.
  Interventions: Other: Test Product G
- Test Product H (Experimental): After irradiation of the test area with a sun simulator with an increment of UV radiation of 1.25, test product will be applied. The dose of test product will be measured in accordance to the application volume (2 mg/cm^2 (± 0.05 mg/cm^2) and it will be applied using a micro litre syringe in approximately 15-30 small droplets all over the test area. Test product will be then quickly spread by gently rubbing with a non-saturated finger cot, first with rotating followed by crosswise movements for a final uniform coating on the skin. Spreading time will be between 20 and 50 s. After waiting for 15 to 30 min, the test area will be again irradiated (increment of 1.12 or 1.25) with the sun simulator. The irradiation time will depend on the expected SPF of the test product, participants' skin prototype, determined MED after irradiation and actual power of sun simulator.
  Interventions: Other: Test Product H

INTERVENTIONS:
Other: Negative Control — Untreated area
  Arms: Negative Control
Other: Positive Control — High SPF Standard P3/SPF 15
  Arms: Positive Control
Other: Test Product A — Yosemite Falls (Forte Day SPF upgrade) Variant A
  Arms: Test Product A
Other: Test Product B — Yosemite Falls (Forte Day SPF upgrade) Variant B
  Arms: Test Product B
Other: Test Product C — Yosemite Falls (Forte Day SPF upgrade) Variant C
  Arms: Test Product C
Other: Test Product D — Yosemite Falls (Forte Day SPF upgrade) Variant D
  Arms: Test Product D
Other: Test Product E — Yosemite Falls (Forte Day SPF upgrade) Variant E
  Arms: Test Product E
Other: Test Product F — Yosemite Falls (Forte Day SPF upgrade) Variant F
  Arms: Test Product F
Other: Test Product G — Yosemite Falls (Forte Day SPF upgrade) Variant G
  Arms: Test Product G
Other: Test Product H — Yosemite Falls (Forte Day SPF upgrade) Variant H
  Arms: Test Product H

SUMMARY:
The study aims to determine the Sun Protection Factor (SPF) of 8 cosmetic products in vivo on the back of human participants, according to the International Standard Sun Protection Test method by using a sun simulator.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the study and willingness to participate as demonstrated by voluntary written informed consent
* Age between 18 to 70 years (inclusive)
* Uniform skin and no erythema or dark pigmentation in the test area
* Skin type I, II or III according to Fitzpatrick scale
* Individual typological angle (ITA°) > 28 in the test area
* Willingness to discontinue the use of detergents, cosmetic products in the treatment areas and to avoid any exposure of the test area to artificial or natural ultraviolet (UV) light throughout the study

Exclusion Criteria:

* Breast feeding, pregnant women or who are intending to become pregnant over study duration
* Acquired immunodeficiency syndrome (AIDS) or infectious hepatitis, insulin dependent diabetes, cancer, active skin disease at the test area, asthma or hypertension if not medicated, medical history of dysplastic nevi or melanoma, allergies to cosmetic products
* Electronic implant that cannot be removed during irradiation
* Sun exposition, UV therapy, artificial tanning within the last 4 weeks, or irregularly tanned skin in the test area
* Application of leave-on cosmetics at the test area within the last 24 h prior to the study start
* Moles, tattoos, scars, irritated skin, hair, etc. at the test area that could influence the investigation
* Usage of medications with known photo-toxic and/or photo-sensitizing potential within the last 14 days prior to study start and/or throughout the entire study course
* Systemic therapy with immuno-suppresive drugs and/or antihistamines within last 7 days prior to study start and/or throughout the entire study course
* Systemic therapy with anti-phlogistic agents or analgetics within last 3 days prior to study start and/or throughout the entire study course
* Participation or in waiting period of 2 months after participation in similar cosmetic and/or pharmaceutical UV studies
* Known or suspected intolerance or hypersensitivity to cosmetic products
* Alcohol or other substance of abuse within the last 5 years
* Employee of the sponsor or the study site or members of their immediate family

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Visual evaluation of irradiated skin | Upto 2 weeks
  Visual evaluation of irradiated test area will be carried out to determine Minimal Erthemal Dose (MED). The lowest irradiation dose producing perceptible erythema will be chosen as MED. The individual SPF (SPFi) for each test product will be determined by calculating the ratio of the MED on test product protected skin (MEDp) to the MED on unprotected skin (MEDu).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Schenefeld, Schleswig-Holstein, Germany